CLINICAL TRIAL: NCT00487604
Title: Retrospective Study of the Impact of Drug Eluting Stents on Intermediate Term Survival, Cardiovascular Outcomes Including Revascularization, Bleeding Rates and Economic Costs
Brief Title: Retrospective Study of the Impact of Drug Eluting Stents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Providence Health & Services (Other)
Other Study IDs: PMRC1371
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug Eluting Stent; Bare Metal Stent; Subacute thrombosis; Bleeding; Economic
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether the use of drug eluting stents is associated with higher rates of death, myocardial infarction, and major bleeding. In addition, the overall economic costs of implanting drug eluting stents compared to bare metal stents will be assessed.

DETAILED DESCRIPTION:
A major limitation of percutaneous coronary stenting compared to coronary artery bypass grafting surgery has been the significantly higher need for repeat revascularization due to restenosis occurring at or near the stent site. By eluting a potent anti-proliferative agent from a polymer coated stent in a time-controlled manner, it has been possible to markedly inhibit intimal proliferation that results from implantation of a bare metal stent, dramatically reducing the need for future target lesion revascularization.

Recent angioscopic and autopsy studies have demonstrated markedly delayed and incomplete endothelialization following drug-eluting stent implantation. These events are rarely observed following bare metal stent implantation. In addition, drug-eluting stents have been associated with hypersensitivity reactions, which may predispose patients to subacute thrombosis. Finally, serial intra-coronary ultrasound studies demonstrate late stent mal-apposition, which is believed to create a possible nidus for thrombus formation.

By means of examining several extensive administrative databases, this study will retrospectively examine approximately 9,800 consecutive patients who underwent either bare metal or drug eluting coronary artery stenting at Sacred Heart Medical Center, Spokane, WA between March 1, 2001 and March 30, 2006. Time frame of follow-up is at least 18 months.

Comparison: The strategy of implanting stents during three time periods will be compared to each other. In the first study period which occurred prior to commercial release of the Cypher drug eluting stent, all patients received bare metal stents. The second study group will include all patients from the time frame between release of the Cypher stent and the Taxus drug eluting stent (approximately one year) after which a contractual decision was made to only utilize Taxus stents. During second time frame of corresponding to availability of the Cypher stent, about 30% of total stent cases received drug eluting stents predominately for "on label" indications. The third study group occurred during a time-frame when Taxus drug eluting stents were implanted in about 90% of overall patients including many with "off label" indications.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery stenting between March 1, 2001 and March 30, 2006

Exclusion Criteria:

* Implanted investigational drug eluting stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9800 (Estimated)
Dates: Start 2007-05; Study Completion 2008-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Ring, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Sacred Heart Medical Center, Spokane, Washington, United States